CLINICAL TRIAL: NCT06839989
Title: The Mpox Biology, Outcome, Transmission and Epidemiology Project - HIV Immunization and Vaccination Against Mpox eXposure Trial
Brief Title: An Immunogenicity and Safety Trial of MVA-BN in Adults Living With HIV for the Prevention of Mpox Infection, in Kinshasa, DRC
Acronym: Mbote-HIVAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: MSF Médecins Sans Frontières Belgium (Unknown); Institut National pour la Recherche Biomedicale (INRB) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mbote-HIVAX
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Mpox (Monkeypox)
Keywords: MVA-BN; Vaccination; Mpox
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CD4 <200 (Experimental): Participants in this arm are stratified in the group with participants with a CD4 level below 200cells/µL.
  Interventions: Biological: Mpox vaccination with MVA-BN
- CD4 200-499 (Experimental): Participants in this arm are stratified in the group with participants with a CD4 level between 200 and 499 cells/µL.
  Interventions: Biological: Mpox vaccination with MVA-BN
- CD4 >= 500 (Experimental): Participants in this arm are stratified in the group with participants with a CD4 level of 500cells/µL or more.
  Interventions: Biological: Mpox vaccination with MVA-BN

INTERVENTIONS:
Biological: Mpox vaccination with MVA-BN — All participants will be vaccinated on day 0 with the MVA-BN vaccine followed by a second injection on day 28.

SUMMARY:
This is an open-label, phase 2, immunogenicity and safety trial of the MVA-BN vaccine for the prevention of mpox in adults living with HIV with different level of CD4 counts in Kinshasa, DRC.

The study team aims to investigate whether the administration of 2 standard subcutaneous doses of the Modified Vaccinia Ankara of Bavarian Nordic (MVA-BN) vaccine given 28 days apart, is immunogenic and safe when administered to People Living with HIV (PLHIV) with different levels of CD4 counts in the Democratic Republic of the Congo (DRC).

Enrollment will be stratified according to three different subgroups based on CD4 counts assessed during visit 1A: <200 cells/µL; 200 to 499 cells/µL; ≥ 500 cells/µL. A total of 600 participants will be included in the trial, with 200 participants per subgroup.

All participants will be invited to 6 trial visits over a period of 7 months.

This study will take place in cooperation with the National Programme for the Fight against AIDS (PNLS), the 'Programme Elargi de Vaccination (PEV)' and the 'Institut National de Santé Publique (INSP)'. As part of the response to the current mpox epidemic in DRC, a large cohort of about 10,000 individuals living in Kinshasa will be vaccinated in this program. Vaccination will take place in the Centre Hospitalier Kabinda (CHK) and the Pakadjuma Health Centre. All people living with HIV (PLHIV) with the intention to be vaccinated in the CHK, will be asked for their willingness to participate in the MBOTE-HIVAX clinical trial until the sample size of 600 participants needed for this clinical trial is reached.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 45 years at time of informed consent
* Able and willing to provide written informed consent
* Infected with HIV and receiving combination antiretroviral therapy (ART) for ≥ 8 weeks prior to study entry and vaccination
* Preparedness to follow the study schedule
* Willingness to use contraception for 1 month after each vaccination (only for women of childbearing potential)

Exclusion Criteria:

* A known history of mpox and/or smallpox
* A known history of vaccination with 1st, 2nd or 3rd generation smallpox vaccines, or vaccine platforms that contain MVA as a vector
* Planned MVA-based vaccination (other than study vaccination) during the trial
* Close contact to a confirmed mpox case in the 3 weeks prior to study enrollment
* Uncontrolled severe infection or other condition requiring hospitalization
* Pregnancy
* History of anaphylaxis or severe allergic reaction to any vaccine or known allergy to one of the components of the study vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rates for monkeypox virus (MPXV) neutralizing antibodies | 2 weeks after the last vaccine dose
  Seroconversion two weeks after administration of two standard doses of MVA-BN, defined as either the appearance of an MPXV neutralizing antibody titre (NT50) greater than or equal to the detection limit for initially seronegative participants or more than doubling of the antibody titre compared to baseline for participants seropositive at baseline

SECONDARY OUTCOMES:
Safety and reactogenicity of the MVA-BN vaccine in PLHIV | Up to day 14 and until end of participation
  Solicited local AEs (pain, redness, swelling, induration, and itch at the injection site) and systemic AEs (generalized myalgia, headache, fatigue, nausea and/or vomiting, chills and/or fever (≥ 38.0°C)) up to day 14 post vaccination
  Unsolicited AEs up to day 14 post vaccination
  SAEs until the end of participation
Seroconversion rates for vaccinia virus (VACV) neutralizing antibodies | 2 weeks after last vaccine dose
  Seroconversion two weeks after administration of two standard doses of MVA-BN, defined as either the appearance of an VACV neutralizing antibody titre (NT50) greater than or equal to the detection limit for initially seronegative participants or more than doubling of the antibody titre compared to baseline for participants seropositive at baseline.
Waning of MPXV neutralizing antibodies in PLHIV | On day 14 and month 6
  The ratio between neutralizing antibody titre against MPXV at 6 months (D28 + 6M) versus 14 days (D28 + 14 days) after administration of two standard doses of MVA-BN.
Waning of VACV neutralizing antibodies in PLHIV | On day 14 and month 6
  The ratio between neutralizing antibody titre against VACV at 6 months (D28 + 6M) versus 14 days (D28 + 14 days) after administration of two standard doses of MVA-BN.
Seroconversion rates and IgG antibody titre dynamics against MPXV and VACV antigens in serum | day 0 (prior to first dose), Day14, Day 28, Day 28+14 days, Day 28+6Months
  The absolute IgG antibody titre against the following antigens: A35R, H3L, B2R, A5L, A27L, B6R, E8L and A29L from mpox, and A33R and B5 from vaccinia virus at D14, D28 (second dose), D28+14d, D28+6M after administration of two standard doses of MVA-BN, be defined as either the appearance of Median Fluorescent Values (MFI) greater than the detection limit for initially seronegative participants or more than doubling of the antibody titre compared to baseline for participants seropositive at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Liesenborghs, MD, Principal Investigator — Institute of Tropical Medicine
Locations (1):
- Centre Hospitalier Kabinda, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR